CLINICAL TRIAL: NCT07319819
Title: The Effectiveness of Case-Based Educational Scenarios in the Metaverse Environment on Enhancing Interpersonal Communication Skills, Path of Academic Engagement, and Reducing Mind-Wandering in University Nursing Students
Brief Title: Effectiveness of Case-Based Educational Scenarios in the Metaverse on Interpersonal Communication Skills, Academic Engagement, and Mind-Wandering in University Nursing Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Port Said University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SCBR-449
Record Dates: First submitted 2025-12-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-03

CONDITIONS: Communication
MeSH Terms: conditions — Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metaverse Case-Based Scenario Group (Experimental): Participants in this arm will receive case-based educational scenarios delivered through a metaverse environment as part of their psychiatric nursing coursework. Students will engage in interactive virtual simulations with virtual patients and healthcare teams to practice interpersonal communication in complex, emotionally charged psychiatric scenarios.
  Interventions: Behavioral: Metaverse Case-Based Educational Scenarios
- Control (No Intervention): Participants in this arm will receive the usual psychiatric nursing teaching methods without exposure to metaverse-based case scenarios. They will continue to follow the standard curriculum delivered through conventional classroom or existing e-learning formats.

INTERVENTIONS:
Behavioral: Metaverse Case-Based Educational Scenarios — The intervention consists of structured case-based scenarios delivered via an immersive metaverse platform, where students interact in real time with virtual patients and peers. Sessions will be designed to promote interpersonal communication, empathy, and academic engagement and to reduce mind-wandering during psychiatric nursing education activities. (You may later specify number of sessions, duration per session, and total intervention period when finalized.)
  Arms: Metaverse Case-Based Scenario Group

SUMMARY:
This randomized controlled trial will evaluate the effect of case-based educational scenarios delivered in a metaverse environment on interpersonal communication skills, academic engagement, and mind-wandering among undergraduate nursing students. Fourth-level nursing students will be randomly assigned either to metaverse-based case scenarios integrated into their psychiatric nursing education or to usual teaching without metaverse exposure. Outcomes will be measured using validated scales for interpersonal communication, learning engagement, and mind-wandering before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

Registered undergraduate nursing students at the Faculty of XXX University, XXX.

Enrolled in the 4th level of the nursing program in the academic year 2024-2025.

Able and willing to provide informed consent to participate.

Exclusion Criteria:

Students not registered in the 4th level during the study period. Students who previously completed formal metaverse-based psychiatric nursing training (if applicable).

Students unwilling to participate or who withdraw consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Interpersonal Communication Skills Score | Baseline (pre-intervention) and immediately post-intervention (end of teaching period)
  Total score on the Interpersonal Communication Skills tool assessing communication abilities in clinical and academic interactions

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schaufeli WB, Martínez IM, Pinto AM, Salanova M, Bakker AB. Burnout and engagement in university students: A cross-national study. J Cross Cult Psychol. 2002;33(5):464-481.
- [Background] Li, X.Y.; Huang, R. The Revision report of the University Student Learning Engagement Scale (UWES-S). Psychol. Res. 2010, 3, 84-88